CLINICAL TRIAL: NCT04527549
Title: The BAMM2 (BRAF, Autophagy, MEK Inhibition in Melanoma) Study: A Randomized Double Blind Phase II Study of Dabrafenib and Trametinib With or Without Hydroxychloroquine in Advanced BRAF V600E/K Melanoma With Elevated LDH
Brief Title: Testing Dabrafenib and Trametinib With or Without Hydroxychloroquine in Stage IIIC or IV BRAF V600E/K Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EA6191; NCI-2020-04552 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EA6191 (Other: ECOG-ACRIN Cancer Research Group); EA6191 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2020-08-24; First posted 2020-08-26 (Actual); Results first posted 2024-08-22 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Clinical Stage IV Cutaneous Melanoma AJCC v8; Locally Advanced Melanoma; Pathologic Stage IIIC Cutaneous Melanoma AJCC v8; Pathologic Stage IV Cutaneous Melanoma AJCC v8; Unresectable Melanoma
MeSH Terms: interventions — dabrafenib; Hydroxychloroquine; trametinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (dabrafenib, trametinib, hydroxychloroquine) (Experimental): Patients receive dabrafenib mesylate PO BID, trametinib dimethyl sulfoxide PO QD, and hydroxychloroquine sulfate PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dabrafenib mesylate; Drug: Hydroxychloroquine; Drug: Trametinib dimethyl sulfoxide
- Arm B (dabrafenib, trametinib, placebo) (Active Comparator): Patients receive dabrafenib mesylate PO BID, trametinib dimethyl sulfoxide PO QD, and placebo PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dabrafenib mesylate; Drug: Placebo Administration; Drug: Trametinib dimethyl sulfoxide

INTERVENTIONS:
Drug: Dabrafenib mesylate — Given PO
  Other Names: NSC 763760; GSK2118436A (free base); Tafinlar®; GSK2118436B
Drug: Hydroxychloroquine — Given PO
  Other Names: Hydroxychloroquine sulfate; Plaquenil
  Arms: Arm A (dabrafenib, trametinib, hydroxychloroquine)
Drug: Placebo Administration — Given PO
  Arms: Arm B (dabrafenib, trametinib, placebo)
Drug: Trametinib dimethyl sulfoxide — Given PO
  Other Names: trametinib; GSK1120212B; TMT212-NXA; JTP-74057; JTP-78296; JTP-75303; Mekinist®; NSC 763093

SUMMARY:
This phase II trial investigates how well adding hydroxychloroquine to the standard treatment of dabrafenib and trametinib works to overcome resistance and delay disease progression in treating patients with stage IIIC or IV BRAF V600E/K melanoma. Hydroxychloroquine may cause cell death in tumor cells that rely on a process called "autophagy" for survival. Dabrafenib and trametinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving hydroxychloroquine together with dabrafenib and trametinib may work better than dabrafenib and trametinib alone to shrink and stabilize the cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the rate of one year progression-free survival (PFS) when hydroxychloroquine sulfate (hydroxychloroquine) or placebo is added to dabrafenib mesylate (dabrafenib) and trametinib dimethyl sulfoxide (trametinib) in advanced BRAFV600E/K melanoma with elevated lactate dehydrogenase (LDH).

SECONDARY OBJECTIVES:

I. To compare the PFS of both arms. II. To evaluate the best overall response rate by treatment arm. III. To evaluate the complete response (CR) rate by treatment arm. IV. To evaluate the adverse event rate by treatment arm. V. To evaluate overall survival (OS) by treatment arm.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive dabrafenib mesylate orally (PO) twice daily (BID), trametinib dimethyl sulfoxide PO once daily (QD), and hydroxychloroquine sulfate PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive dabrafenib mesylate PO BID, trametinib dimethyl sulfoxide PO QD, and placebo PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have locally advanced unresectable stage IIIC or stage IV melanoma
* Patient must have BRAF V600E or BRAF V600K tumor genotype based on a Clinical Laboratory Improvement Act (CLIA) approved assay
* Patient must have serum LDH > Upper limit of normal per institution standards
* Patient must have measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Baseline measurements of sites of disease must be obtained within 3 weeks prior to study randomization
* Patient must have been treated with prior immune checkpoint inhibitor therapy (anti PD-1 antibody, anti-CTLA-4 antibody or a combination regimen including either or both agents) either in the adjuvant or metastatic setting. Patient may have received investigational agents in combination with standard therapy, as long as it was adhering to the timeframes below

  * Patient must have discontinued active immunotherapy (IL-2, interferon, anti-CTLA-4 antibody, anti-PD-1 antibody etc.) or chemotherapy at least 4 weeks prior to randomization
  * Patient must have discontinued any oral targeted therapy at least 2 weeks prior to randomization
* Patient may have been treated with prior adjuvant therapy including combined BRAF and MEK inhibitor therapy. Patients will be eligible if they tolerated this therapy and did not discontinue the therapy due to toxicity AND >= 6 months have elapsed since the end of adjuvant BRAF and MEK inhibition.
* Patient may have been treated with prior chemotherapy or radiation therapy
* Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* All females of childbearing potential must have a blood test or urine study within 14 days prior to randomization to rule out pregnancy.
* Women of childbearing potential and sexually active males must not expect to conceive or father children by using accepted and effective method(s) of contraception or abstaining from sexual intercourse for the duration of their participation in the study and for 4 months after the last dose of protocol treatment
* Patient must have recovered from clinically significant reversible toxicities from previous treatment prior to randomization. Abnormal laboratory values may be grade 1, as long as they meet the eligibility criteria for organ and marrow function
* Patient must be able to swallow and retain oral medication and must not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels
* Patient must have the ability to understand and the willingness to sign a written informed consent document. Patients with impaired decision-making capacity (IDMC) who have a legally authorized representative (LAR) or caregiver and/or family member available will also be considered eligible
* Absolute neutrophil count >= 1,500/mcL (obtained =< 14 days prior to protocol randomization)
* Platelets >= 100,000/mcL (obtained =< 14 days prior to protocol randomization)
* Total bilirubin =< institutional upper limit of normal (ULN) (obtained =< 14 days prior to protocol randomization)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3.0 x institutional ULN (obtained =< 14 days prior to protocol randomization)
* Creatinine =< 1.5 x institutional ULN (obtained =< 14 days prior to protocol randomization)
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patient with asymptomatic new or progressive brain metastases (active brain metastases) are eligible if the treating physician determines that CNS specific treatment is not required

  * NOTE: Patient with treated brain metastases are eligible. No brain imaging is required, however, 1 week must elapse after gamma knife therapy. Patient treated with whole brain radiation that have been stable for 2 months are eligible. Patient are excluded if they have leptomeningeal disease or metastases causing spinal cord compression that are symptomatic or untreated or not stable (documented by imaging) for at least 3 months or requiring corticosteroids. Patients on a stable dose of corticosteroids for at least 1 month or who have been off of corticosteroids for at least 1 week are eligible

Exclusion Criteria:

* Receiving any other investigational anticancer therapy during the period on study or the 4 weeks prior to randomization
* Patients received BRAF and MEK inhibitor therapy in the metastatic setting
* Patients who are experiencing an objective partial response to immunotherapy at the time of study enrollment
* Pregnant or breast-feeding; due to the potential harm to an unborn fetus and possible risk for adverse events in nursing infants with the treatment regimens being used. A female of childbearing potential is defined as any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy; or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* A history of interstitial lung disease (ILD) or chronic pneumonitis

  * NOTE: If there is radiographic evidence of ILD that is clinically insignificant and asymptomatic, the patient would be eligible
* Porphyria or psoriasis due to risk of disease exacerbation unless the disease is well controlled and they are under the care of a specialist for the disorder who agrees to monitor the patient for exacerbations
* Previously documented retinal vein occlusion
* A history or evidence of increased cardiovascular risk including:

  * Left ventricular ejection fraction (LVEF) < institutional lower limit of normal measured within 14 days prior to randomization
  * A QT interval corrected for heart rate using the Bazett's formula >= 480 msec
  * Current clinically significant uncontrolled arrhythmias. Exception: Patients with controlled atrial fibrillation for > 30 days prior to randomization are eligible
  * Acute coronary syndromes (including myocardial infarction and unstable angina), coronary angioplasty, or stenting within 6 months prior to randomization
  * Abnormal cardiac valve morphology (>= grade 2) documented by echocardiogram unless a cardiologist concludes the valve abnormality is not clinically significant. Patients with grade 1 abnormalities (i.e., mild regurgitation/stenosis) are eligible
  * Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* Serious concurrent infection or medical illness, including psychiatric disorders, which would jeopardize the ability of the patient to receive the treatment outlined in this protocol with reasonable safety
* Receiving concurrent therapy for their tumor (i.e. chemotherapeutics or investigational agents). Radiotherapy delivered to palliate pain is allowed as long as it is not targeting a lesion that meets RECIST criteria for progression. Radiation therapy to the surgical bed with gamma knife radiotherapy while on treatment during the first cycle is allowed for small volume surgically resected brain metastases. Gamma knife radiotherapy for known active, asymptomatic small volume central nervous system (CNS) lesions may be performed during the first cycle while on study. Radiotherapy for new CNS lesions identified beyond the first cycle is not allowed on study
* Immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to study drug, or excipients or to dimethyl sulfoxide (DMSO)
* Prior cytochrome P450 enzyme -inducing anticonvulsant drugs (extended-interval aminoglycoside dosing [EIADs]) (i.e. phenytoin, carbamazepine, phenobarbital, primidone or oxcarbazepine) within 4 weeks prior to randomization
* Current use of a prohibited medication described in the protocol due to potential drug-drug interaction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-01-08 (Actual); Study Completion 2024-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Amaravadi, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (199):
- United States (199):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Saint Francis Cancer Center, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Beebe South Coastal Health Campus, Frankford, Delaware
  - Beebe Medical Center, Lewes, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - UM Sylvester Comprehensive Cancer Center at Aventura, Aventura, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Saint Anthony's Health, Alton, Illinois
  - Rush - Copley Medical Center, Aurora, Illinois
  - Loyola Center for Health at Burr Ridge, Burr Ridge, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Loyola Medicine Homer Glen, Homer Glen, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Marjorie Weinberg Cancer Center at Loyola-Gottlieb, Melrose Park, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Reid Health, Richmond, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic PC - Ames, Ames, Iowa
  - McFarland Clinic PC-Boone, Boone, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Mission Cancer and Blood - Laurel, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - McFarland Clinic PC-Trinity Cancer Center, Fort Dodge, Iowa
  - Trinity Regional Medical Center, Fort Dodge, Iowa
  - McFarland Clinic PC-Jefferson, Jefferson, Iowa
  - McFarland Clinic PC-Marshalltown, Marshalltown, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Saint Elizabeth Boardman Hospital, Boardman, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC-Miami Valley Hospital North, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Dayton Physicians LLC-Upper Valley, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Joseph Warren Hospital, Warren, Ohio
  - Saint Elizabeth Youngstown Hospital, Youngstown, Ohio
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Marshfield Clinic - Ladysmith Center, Ladysmith, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be made available upon request as per the ECOG-ACRIN Data Sharing Policy.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was activated on October 23, 2020, and closed to accrual on March 1, 2023 due to slower than expected accrual. The first patient was enrolled on June 1st, 2021.
Period: Overall Study
Arm/Group | Arm A (Dabrafenib, Trametinib, Hydroxychloroquine) | Arm B (Dabrafenib, Trametinib, Placebo)
Started | 3 | 2
Completed | 2 | 1
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Dabrafenib, Trametinib, Hydroxychloroquine) | Arm B (Dabrafenib, Trametinib, Placebo) | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Continuous [Median (Full Range); unit: years] | 38 [30 to 61] | 68 [64 to 72] | 61 [30 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: One-year Progression-free Survival Rate
Description: Progression-free survival is defined as the time from randomization to progression or death, whichever occurs first. Progression is defined as appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions, or at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
  One-year progression-free survival rate is estimated from the Kaplan-Meier progression-free survival curve.
Time Frame: Assessed every 2 months until 6 months after completion of study treatment, up to 1 year
Population: Only patients who received treatment were included in the analysis.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (Dabrafenib, Trametinib, Hydroxychloroquine) | Arm B (Dabrafenib, Trametinib, Placebo)
Number analyzed (Participants) | 2 | 2
proportion of participants | 0.5 [0.006 to 0.91] | NA [NA to NA] — 1-year PFS rate could not be estimated as one patient experienced progression within 1 year and the other patient withdrew consent prior to 1 year.

2. Secondary Outcome: Progression-free Survival
Description: Progression-free survival is defined as the time from randomization to progression or death, whichever occurs first. Progression is defined as appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions, or at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: Assessed every 2 months until 6 months after completion of study treatment, up to 3 years
Population: Only patients received treatment were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Dabrafenib, Trametinib, Hydroxychloroquine) | Arm B (Dabrafenib, Trametinib, Placebo)
Number analyzed (Participants) | 2 | 2
months | 12.5 [7 to 18] | NA [2 to NA] — Median was not reached. The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

3. Secondary Outcome: Proportion of Patients With Best Overall Response
Description: Best overall response is defined as either complete response or partial response.
  Complete response is defined as disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial response is defined as persistence of one or more non-target lesion(s) and at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Assessed every 2 months until 6 months after completion of study treatment, up to 3 years
Population: Only patients received treatment were included in the analysis.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (Dabrafenib, Trametinib, Hydroxychloroquine) | Arm B (Dabrafenib, Trametinib, Placebo)
Number analyzed (Participants) | 2 | 2
proportion of participants | 1.0 [0.16 to 1.00] | 0.5 [0.01 to 0.99]

4. Secondary Outcome: Proportion of Patients With Complete Response
Description: Complete response is defined as disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
Time Frame: Assessed every 2 months until 6 months after completion of study treatment, up to 3 years
Population: Only patients received treatment were included in the analysis.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (Dabrafenib, Trametinib, Hydroxychloroquine) | Arm B (Dabrafenib, Trametinib, Placebo)
Number analyzed (Participants) | 2 | 2
proportion of participants | 0 [0 to 0.84] | 0 [0 to 0.84]

5. Secondary Outcome: Adverse Event Rate
Description: Proportion of patients with treatment-related adverse events of grade 3 or higher.
Time Frame: Assessed every 4 weeks while on treatment and for 30 days after the end of treatment, up to 3 years
Population: Only patients who received treatment were included in this analysis.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (Dabrafenib, Trametinib, Hydroxychloroquine) | Arm B (Dabrafenib, Trametinib, Placebo)
Number analyzed (Participants) | 2 | 2
proportion of participants | 0.5 [0.01 to 0.99] | 0.5 [0.01 to 0.99]

6. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from randomization to death or date last known alive.
Time Frame: Assessed every 2 months until 6 months after completion of study treatment, up to 3 years
Population: Only patients received treatment were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Dabrafenib, Trametinib, Hydroxychloroquine) | Arm B (Dabrafenib, Trametinib, Placebo)
Number analyzed (Participants) | 2 | 2
months | NA [NA to NA] — Median was not reached. The lower and upper limit of the 95% confidence interval were not calculable because an insufficient number of participants reached the event at the final time point for assessment. | NA [2 to NA] — Median was not reached. The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

ADVERSE EVENTS:
Time Frame: Assessed every 4 weeks while on treatment and for 30 days after the end of treatment, up to 3 years
Description: Only patients who received treatment are included in this analysis.
Arm/Group | Arm A (Dabrafenib, Trametinib, Hydroxychloroquine) | Arm B (Dabrafenib, Trametinib, Placebo)
All-Cause Mortality (participants affected / at risk) | 0/2 | 1/2
Serious Adverse Events (participants affected / at risk) | 1/2 | 1/2
Other Adverse Events (participants affected / at risk) | 2/2 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Dabrafenib, Trametinib, Hydroxychloroquine) (N=2) | Arm B (Dabrafenib, Trametinib, Placebo) (N=2)
Fever (General disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Arterial thromboembolism (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Dabrafenib, Trametinib, Hydroxychloroquine) (N=2) | Arm B (Dabrafenib, Trametinib, Placebo) (N=2)
Anemia (Blood and lymphatic system disorders) | 2 | 0
Chills (General disorders) | 2 | 1
Fatigue (General disorders) | 2 | 1
Fever (General disorders) | 2 | 0
Flu like symptoms (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
General disorders and administration site conditions - Other, specify (General disorders) | 1 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 0
Mucositis oral (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Bruising (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Alkaline phosphatase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Weight loss (Investigations) | 1 | 0
White blood cell decreased (Investigations) | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0
Investigations - Other, specify (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Hyperlipidemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Extrapyramidal disorder (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 1
Vasovagal reaction (Nervous system disorders) | 0 | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 0 | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dry eye (Eye disorders) | 1 | 0
Eye disorders - Other, specify (Eye disorders) | 1 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Urinary urgency (Renal and urinary disorders) | 1 | 0
Flushing (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-19): https://cdn.clinicaltrials.gov/large-docs/49/NCT04527549/Prot_SAP_000.pdf